CLINICAL TRIAL: NCT04196088
Title: AIDA: A Multicenter, Prospective, Randomized Controlled Trial to Evaluate the Clinical Efficacy and Safety of Artificial Intelligence (AI) Detection of Adenomas (AIDA) With Standard High Definition With Light in Screening Colonoscopy
Brief Title: To Compare Artificial Intelligence Software Aided Adenoma Detection in Screening Colonoscopies Versus Standard Colonoscopy Without Artificial Intelligence Software Assistance in Participants Between 45 and 75 Years of Age
Acronym: AIDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Docbot, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Docbot AIDA: Ultivision_002
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Adenoma; Colorectal Polyp; Colorectal Adenocarcinoma; Colorectal SSA
Keywords: screening colonoscopy; artificial intelligence; software as a medical device; adenoma detection rate; adenomas per endoscopy; mean adenomas per colonoscopy; colorectal cancer; medical device
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Triple (Participant, Pathologist, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Ultivision AI Software enhanced screening colonoscopy (Active Comparator): Ultivision Artificial Intelligence enhanced screening colonoscopies will be performed.
  Interventions: Device: Ultivision Artificial Intelligence Software
- No AI enhancement screening colonoscopy (Placebo Comparator): Screening colonoscopies without Artificial Intelligence enhancement will be performed.
  Interventions: Device: No Artificial Intelligence Software enhancement

INTERVENTIONS:
Device: Ultivision Artificial Intelligence Software — Screening Colonoscopy
  Arms: Ultivision AI Software enhanced screening colonoscopy
Device: No Artificial Intelligence Software enhancement — Screening Colonoscopy
  Arms: No AI enhancement screening colonoscopy

SUMMARY:
The aim of this study is to assess the efficacy of Ultivision Artificial Intelligence (AI) Software in detecting adenomas in screening colonoscopy procedures. The safety of Ultivision AI Software will also be assessed. A subset of the subjects will enter a roll-in period for clinical trial safety assessment. The remainder of subjects who are eligible will enter the detection phase which comprises a screening colonoscopy procedure. In the detection phase, subjects will be randomized to a screening colonoscopy with Ultivision AI Software enhancement or without AI Software enhancement. The study will measure the mean adenomas per colonoscopy procedure, as defined by the protocol, detected while receiving either treatment option.

ELIGIBILITY:
Primary Inclusion Criteria.

1. Average risk asymptomatic subjects undergoing a first colonoscopy (screening) or screening colonoscopy at least 10 years after prior colonoscopy.
2. Aged 45 years to aged 75 years at the time of enrollment.
3. Capable of providing written informed consent and willing and able to adhere to all protocol requirements, and/or the subject's legally acceptable representative(s) capable of providing written informed consent.

Primary Exclusion Criteria.

1. History of any colorectal cancer or colon adenomas.
2. History of inflammatory bowel disease, including Crohn's disease or ulcerative colitis.
3. Family history of colon cancer or precancerous colon polyp in a first degree relative before age 50.
4. Polyposis syndromes including Familial Adenomatous Polyposis, Cowden syndrome, Lynch syndrome, Peutz-Jeghers syndrome, MUTYH Associated Polyposis, Familial Colorectal Cancer Type X.
5. Surveillance, therapeutic, preoperative, or diagnostic colonoscopy.
6. Colonoscopy for work-up of abdominal or pelvic symptoms including abdominal pain, flank pain, pelvic pain, subject report of altered stool, subject report of anemia within the past 12 months, subject report of gastrointestinal bleeding including bright red blood per rectum or tarry stools, constipation, diarrhea, subject reported history of abdominal or pelvic mass, subject report of unintentional weight loss.
7. Workup or referral to diagnose or evaluate abnormal imaging of the abdomen or pelvis.
8. Positive Fecal Immunochemical Test history.
9. Severe co-mobordity, including end-stage cardiovascular, pulmonary, liver, or renal disease.
10. History of colon resection, not including the appendix.
11. Currently receiving a therapy not permitted during the trial, as defined in Section 8.3.
12. Any issue that, in the opinion of the investigator, would render the subject unsuitable for participation in the trial.

Enrolled subjects will be eligible for Post-procedure Periods if their colonoscopy meets the following criteria:

1. Adequate bowel preparation score per the Boston Bowel Preparation Scoring System (BBPS) > or equal to 2 in all colonic segments.
2. Colonoscopies with successful cecal intubation.
3. Colonoscopies with withdrawal times of at least 6 minutes.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 978 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Overall adenoma detection, as defined by the protocol, using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  The primary efficacy endpoint is the mean adenomas per colonoscopy procedure (MAP) detection, as defined by the protocol, with Ultivision AI software enhancement to screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI.
Overall adenomas per extraction, as defined by the protocol, using Ultivision AI software in subjects undergoing screening standard hiigh definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  The primary safety endpoint is the adenomas per extraction per colonoscopy procedure (APE), as defined by the protocol, using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus SHDWLC without AI.

SECONDARY OUTCOMES:
Adenoma detection rate, as defined by the protocol, using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  The secondary efficacy endpoint is the adenoma detection rate (ADR) defined as the ratio of screening colonoscopies with at least one adenoma, as defined by the protocol, detected divided by the total number of screening SHDWLC performed with Ultivision AI versus screening SHDWLC performed without AI.

OTHER OUTCOMES:
Advanced adenoma detection rate (AADR) using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  Advanced adenoma detection rate (AADR) on SHDWLC using AI versus SHDWLC without AI.
Sessile serrated adenoma/polyp (SSA/P) detection rate using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  Sessile serrated adenoma/polyp (SSA/P) detection rate on SHDWLC using AI versus SHDWLC without AI.
Polyp detection rate using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  Polyp detection rate on SHDWLC using AI versus SHDWLC without AI.
Flat versus polypoid lesion detection rate using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  Flat versus polypoid lesion detection rate on SHDWLC AI versus SHDWLC without AI.
Polyp location distribution using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  Polyp location distribution on SHDWLC using AI versus SHDWLC without AI.
Surveillance-irrelevant lesion (SIL) and surveillance-relevant lesion (SRL) detection rate using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  Surveillance-irrelevant lesion (SIL) and surveillance-relevant lesion (SRL) detection rates using SHDWLC AI versus SHDWLC without AI.
Post colonoscopy recommended surveillance follow-up interval using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  Recommended surveillance interval after using SHDWLC AI versus SHDWLC without AI.
Colonoscope withdrawal time using Ultivision AI software in subjects undergoing screening standard high definition white light colonoscopy (SHDWLC) versus screening SHDWLC without AI. | through study completion, an average of 1 year
  Colonoscope withdrawal time using SHDWLC AI versus SHDWLC without AI.

CONTACTS AND LOCATIONS:
Overall Officials: Efren Rael, MD, Study Director — Docbot, Inc.
Locations (9):
- United States (9):
  - Gastro Health, Birmingham, Alabama
  - Precision Research Institute, San Diego, California
  - Kansas City Veterans Administration, Kansas City, Kansas
  - Capital Digestive Care, Chevy Chase, Maryland
  - East Side Endoscopy, New York, New York
  - Great Lakes Gastroenterology Research, LLC, Clinical Trials Network, Mentor, Ohio
  - Verity Research Inc., Gastro Health, Fairfax, Virginia
  - Gastrointestinal & Liver Specialists of Tidewater, PLLC, Norfolk, Virginia
  - Wisconsin GI Associates, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zauber AG, Winawer SJ, O'Brien MJ, Lansdorp-Vogelaar I, van Ballegooijen M, Hankey BF, Shi W, Bond JH, Schapiro M, Panish JF, Stewart ET, Waye JD. Colonoscopic polypectomy and long-term prevention of colorectal-cancer deaths. N Engl J Med. 2012 Feb 23;366(8):687-96. doi: 10.1056/NEJMoa1100370. PMID 22356322
- [Background] Brenner H, Chang-Claude J, Seiler CM, Rickert A, Hoffmeister M. Protection from colorectal cancer after colonoscopy: a population-based, case-control study. Ann Intern Med. 2011 Jan 4;154(1):22-30. doi: 10.7326/0003-4819-154-1-201101040-00004. PMID 21200035
- [Background] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Background] Shergill AK, Conners EE, McQuaid KR, Epstein S, Ryan JC, Shah JN, Inadomi J, Somsouk M. Protective association of colonoscopy against proximal and distal colon cancer and patterns in interval cancer. Gastrointest Endosc. 2015 Sep;82(3):529-37.e1. doi: 10.1016/j.gie.2015.01.053. Epub 2015 May 1. PMID 25936449
- [Background] Baxter NN, Goldwasser MA, Paszat LF, Saskin R, Urbach DR, Rabeneck L. Association of colonoscopy and death from colorectal cancer. Ann Intern Med. 2009 Jan 6;150(1):1-8. doi: 10.7326/0003-4819-150-1-200901060-00306. Epub 2008 Dec 15. PMID 19075198
- [Background] Brenner H, Chang-Claude J, Rickert A, Seiler CM, Hoffmeister M. Risk of colorectal cancer after detection and removal of adenomas at colonoscopy: population-based case-control study. J Clin Oncol. 2012 Aug 20;30(24):2969-76. doi: 10.1200/JCO.2011.41.3377. Epub 2012 Jul 23. PMID 22826281
- [Background] Singh H, Nugent Z, Demers AA, Kliewer EV, Mahmud SM, Bernstein CN. The reduction in colorectal cancer mortality after colonoscopy varies by site of the cancer. Gastroenterology. 2010 Oct;139(4):1128-37. doi: 10.1053/j.gastro.2010.06.052. Epub 2010 Jun 20. PMID 20600026
- [Background] Corley DA, Jensen CD, Marks AR, Zhao WK, Lee JK, Doubeni CA, Zauber AG, de Boer J, Fireman BH, Schottinger JE, Quinn VP, Ghai NR, Levin TR, Quesenberry CP. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Apr 3;370(14):1298-306. doi: 10.1056/NEJMoa1309086. PMID 24693890
- [Background] Coe SG, Wallace MB. Assessment of adenoma detection rate benchmarks in women versus men. Gastrointest Endosc. 2013 Apr;77(4):631-5. doi: 10.1016/j.gie.2012.12.001. Epub 2013 Feb 1. PMID 23375528
- [Background] Adler J, Robertson DJ. Interval Colorectal Cancer After Colonoscopy: Exploring Explanations and Solutions. Am J Gastroenterol. 2015 Dec;110(12):1657-64; quiz 1665. doi: 10.1038/ajg.2015.365. Epub 2015 Nov 10. PMID 26553207
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339
- [Background] le Clercq CM, Bouwens MW, Rondagh EJ, Bakker CM, Keulen ET, de Ridder RJ, Winkens B, Masclee AA, Sanduleanu S. Postcolonoscopy colorectal cancers are preventable: a population-based study. Gut. 2014 Jun;63(6):957-63. doi: 10.1136/gutjnl-2013-304880. Epub 2013 Jun 6. PMID 23744612
- [Background] Ahn SB, Han DS, Bae JH, Byun TJ, Kim JP, Eun CS. The Miss Rate for Colorectal Adenoma Determined by Quality-Adjusted, Back-to-Back Colonoscopies. Gut Liver. 2012 Jan;6(1):64-70. doi: 10.5009/gnl.2012.6.1.64. Epub 2012 Jan 12. PMID 22375173
- [Background] van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systematic review. Am J Gastroenterol. 2006 Feb;101(2):343-50. doi: 10.1111/j.1572-0241.2006.00390.x. PMID 16454841
- [Background] Rex DK. Maximizing detection of adenomas and cancers during colonoscopy. Am J Gastroenterol. 2006 Dec;101(12):2866-77. doi: 10.1111/j.1572-0241.2006.00905.x. PMID 17227527
- [Background] Aslanian HR, Shieh FK, Chan FW, Ciarleglio MM, Deng Y, Rogart JN, Jamidar PA, Siddiqui UD. Nurse observation during colonoscopy increases polyp detection: a randomized prospective study. Am J Gastroenterol. 2013 Feb;108(2):166-72. doi: 10.1038/ajg.2012.237. PMID 23381064
- [Background] Lee CK, Park DI, Lee SH, Hwangbo Y, Eun CS, Han DS, Cha JM, Lee BI, Shin JE. Participation by experienced endoscopy nurses increases the detection rate of colon polyps during a screening colonoscopy: a multicenter, prospective, randomized study. Gastrointest Endosc. 2011 Nov;74(5):1094-102. doi: 10.1016/j.gie.2011.06.033. Epub 2011 Sep 1. PMID 21889137
- [Background] Buchner AM, Shahid MW, Heckman MG, Diehl NN, McNeil RB, Cleveland P, Gill KR, Schore A, Ghabril M, Raimondo M, Gross SA, Wallace MB. Trainee participation is associated with increased small adenoma detection. Gastrointest Endosc. 2011 Jun;73(6):1223-31. doi: 10.1016/j.gie.2011.01.060. Epub 2011 Apr 8. PMID 21481861
- [Background] Gralnek IM. Emerging technological advancements in colonoscopy: Third Eye(R) Retroscope(R) and Third Eye(R) Panoramic(TM) , Fuse(R) Full Spectrum Endoscopy(R) colonoscopy platform, Extra-Wide-Angle-View colonoscope, and NaviAid(TM) G-EYE(TM) balloon colonoscope. Dig Endosc. 2015 Jan;27(2):223-31. doi: 10.1111/den.12382. Epub 2014 Nov 17. PMID 25251748
- [Background] Kaminski MF, Hassan C, Bisschops R, Pohl J, Pellise M, Dekker E, Ignjatovic-Wilson A, Hoffman A, Longcroft-Wheaton G, Heresbach D, Dumonceau JM, East JE. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2014 May;46(5):435-49. doi: 10.1055/s-0034-1365348. Epub 2014 Mar 17. PMID 24639382
- [Background] Bisschops R, East JE, Hassan C, Hazewinkel Y, Kaminski MF, Neumann H, Pellise M, Antonelli G, Bustamante Balen M, Coron E, Cortas G, Iacucci M, Yuichi M, Longcroft-Wheaton G, Mouzyka S, Pilonis N, Puig I, van Hooft JE, Dekker E. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Dec;51(12):1155-1179. doi: 10.1055/a-1031-7657. Epub 2019 Nov 11. PMID 31711241
- [Background] Parekh PJ, Oldfield EC 4th, Johnson DA. Bowel preparation for colonoscopy: what is best and necessary for quality? Curr Opin Gastroenterol. 2019 Jan;35(1):51-57. doi: 10.1097/MOG.0000000000000494. PMID 30489414
- [Background] Rex DK, Schoenfeld PS, Cohen J, Pike IM, Adler DG, Fennerty MB, Lieb JG 2nd, Park WG, Rizk MK, Sawhney MS, Shaheen NJ, Wani S, Weinberg DS. Quality indicators for colonoscopy. Am J Gastroenterol. 2015 Jan;110(1):72-90. doi: 10.1038/ajg.2014.385. Epub 2014 Dec 2. No abstract available. PMID 25448873
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Background] Mori Y, Kudo SE, Misawa M, Saito Y, Ikematsu H, Hotta K, Ohtsuka K, Urushibara F, Kataoka S, Ogawa Y, Maeda Y, Takeda K, Nakamura H, Ichimasa K, Kudo T, Hayashi T, Wakamura K, Ishida F, Inoue H, Itoh H, Oda M, Mori K. Real-Time Use of Artificial Intelligence in Identification of Diminutive Polyps During Colonoscopy: A Prospective Study. Ann Intern Med. 2018 Sep 18;169(6):357-366. doi: 10.7326/M18-0249. Epub 2018 Aug 14. PMID 30105375
- [Background] Misawa M, Kudo SE, Mori Y, Cho T, Kataoka S, Yamauchi A, Ogawa Y, Maeda Y, Takeda K, Ichimasa K, Nakamura H, Yagawa Y, Toyoshima N, Ogata N, Kudo T, Hisayuki T, Hayashi T, Wakamura K, Baba T, Ishida F, Itoh H, Roth H, Oda M, Mori K. Artificial Intelligence-Assisted Polyp Detection for Colonoscopy: Initial Experience. Gastroenterology. 2018 Jun;154(8):2027-2029.e3. doi: 10.1053/j.gastro.2018.04.003. Epub 2018 Apr 11. No abstract available. PMID 29653147
- [Background] Delavari A, Salimzadeh H, Bishehsari F, Sobh Rakhshankhah E, Delavari F, Moossavi S, Khosravi P, Nasseri-Moghaddam S, Merat S, Ansari R, Vahedi H, Shahbazkhani B, Saberifiroozi M, Sotoudeh M, Malekzadeh R. Mean Polyp per Patient Is an Accurate and Readily Obtainable Surrogate for Adenoma Detection Rate: Results from an Opportunistic Screening Colonoscopy Program. Middle East J Dig Dis. 2015 Oct;7(4):214-9. PMID 26609349
- [Background] Wang P, Berzin TM, Glissen Brown JR, Bharadwaj S, Becq A, Xiao X, Liu P, Li L, Song Y, Zhang D, Li Y, Xu G, Tu M, Liu X. Real-time automatic detection system increases colonoscopic polyp and adenoma detection rates: a prospective randomised controlled study. Gut. 2019 Oct;68(10):1813-1819. doi: 10.1136/gutjnl-2018-317500. Epub 2019 Feb 27. PMID 30814121
- [Background] Lauby-Secretan B, Vilahur N, Bianchini F, Guha N, Straif K; International Agency for Research on Cancer Handbook Working Group. The IARC Perspective on Colorectal Cancer Screening. N Engl J Med. 2018 May 3;378(18):1734-1740. doi: 10.1056/NEJMsr1714643. Epub 2018 Mar 26. No abstract available. PMID 29580179
- [Background] Zhao S, Wang S, Pan P, Xia T, Chang X, Yang X, Guo L, Meng Q, Yang F, Qian W, Xu Z, Wang Y, Wang Z, Gu L, Wang R, Jia F, Yao J, Li Z, Bai Y. Magnitude, Risk Factors, and Factors Associated With Adenoma Miss Rate of Tandem Colonoscopy: A Systematic Review and Meta-analysis. Gastroenterology. 2019 May;156(6):1661-1674.e11. doi: 10.1053/j.gastro.2019.01.260. Epub 2019 Feb 6. PMID 30738046
- [Background] Rutter CM, Johnson E, Miglioretti DL, Mandelson MT, Inadomi J, Buist DS. Adverse events after screening and follow-up colonoscopy. Cancer Causes Control. 2012 Feb;23(2):289-96. doi: 10.1007/s10552-011-9878-5. Epub 2011 Nov 22. PMID 22105578
- [Background] Levin TR, Zhao W, Conell C, Seeff LC, Manninen DL, Shapiro JA, Schulman J. Complications of colonoscopy in an integrated health care delivery system. Ann Intern Med. 2006 Dec 19;145(12):880-6. doi: 10.7326/0003-4819-145-12-200612190-00004. PMID 17179057
- [Background] Feagins LA, Smith AD, Kim D, Halai A, Duttala S, Chebaa B, Lunsford T, Vizuete J, Mara M, Mascarenhas R, Meghani R, Kundrotas L, Dunbar KB, Cipher DJ, Harford WV, Spechler SJ. Efficacy of Prophylactic Hemoclips in Prevention of Delayed Post-Polypectomy Bleeding in Patients With Large Colonic Polyps. Gastroenterology. 2019 Oct;157(4):967-976.e1. doi: 10.1053/j.gastro.2019.05.003. Epub 2019 May 31. PMID 31158369
- [Background] Sorbi D, Norton I, Conio M, Balm R, Zinsmeister A, Gostout CJ. Postpolypectomy lower GI bleeding: descriptive analysis. Gastrointest Endosc. 2000 Jun;51(6):690-6. doi: 10.1067/mge.2000.105773. PMID 10840301
- [Background] Hwang IK, Shih WJ, De Cani JS. Group sequential designs using a family of type I error probability spending functions. Stat Med. 1990 Dec;9(12):1439-45. doi: 10.1002/sim.4780091207. PMID 2281231